CLINICAL TRIAL: NCT03981263
Title: Study of the Quality of Life in Patients With Standard External Breast Prosthesis Compared to Patients With Custom-made Breast Prosthesis. MEAVANTI Project.
Brief Title: Quality of Life in Patients With Standard External Compared to Custom-made Breast Prosthesis.
Acronym: MEAVANTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RC31/17/0335
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Prospective study; Cross over; Quality of life; Breast; Mastectomy; Breast external prothesis; MEAVANTI prothesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Cross-over (2 periods), prospective, open and monocentric study. The wash-out period will be 15 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MEAVANTI + Standard protheses (Other): The patients will benefit from the experimental prothesis (MEAVANTI), after a wash-out period of 15 days, they will benefit from the standard non-adherent prothesis.
  Interventions: Device: MEAVANTI prothesis; Device: Standard prothesis
- Standard + MEAVANTI protheses (Other): The patients will benefit from the standard non-adherent prothesis, after a wash-out period of 15 days, they will benefit from the experimental prothesis (MEAVANTI).
  Interventions: Device: MEAVANTI prothesis; Device: Standard prothesis

INTERVENTIONS:
Device: MEAVANTI prothesis — The experimental prosthesis is the MEAVANTI prosthesis ("custom-made" non-adherent prosthesis in silicone) which can be calibrated to 5 grams near the breast that remains after a mastectomy to create a visual symmetry but also a weight symmetry.
  This prosthesis takes into account the curve of the breasts and the morphological details such as: skin color of the patients, size of the nipples, height of the nipples, shape of the breast.
  The measurements of the patients will be taken using a 3D scanner (i.e. a scanner that corresponds to a 3d scanning and acquiring device (images), not irradiating), a scale and a colour chart.
Device: Standard prothesis — This prosthesis will be compared with a standard non-adherent prosthesis (class I, silicone and polyurethane film), among the models available in the three ranges of standard prostheses (Amoena, Anita and Thuasne). The brand and model will be left to the patient's choice.

SUMMARY:
Despite improvements in surgical techniques, approximately 30% of mastectomies are still performed. Definitively or temporarily, one of the alternatives to restore a volume in the bra is the external breast prosthesis. The main objective is to evaluate whether the "custom-made" MEAVANTI prosthesis improves the quality of life of patients who have had a mastectomy compared to the external standard prosthesis.

DETAILED DESCRIPTION:
In France, breast cancer is a public health issue with around 59,000 new cases per year. Despite improved surgical techniques, there is still around 30% mastectomy performed every year. Definitively or temporarily, one of the alternatives to restore a volume in the bra is the use of external breast prosthesis. Currently, there are 3 silicone brands that are marketed and refunded. These standard prostheses take into account only the curve of the patients and not the weight of the remaining breast making adaptation difficult to all body types. The difference in breast weights can cause several disorders: postural, pain, discomfort, psychological impact on quality of life as well as medico-economic impact. MEAVANTI is an external breast prosthesis for custom calibration and personalization, which can prevent postural compensation and provide greater comfort.

The main objective of this study is therefore to evaluate whether the MEAVANTI prosthesis improves the quality of life of patients who have undergone a mastectomy compared to the standard prosthesis (through the EORTC questionnaires - European Organization for Research and Treatment of Cancer). This study will be monocentric, cross-over (2 periods), prospective, open with a wash-out period of 15 days. The period of the study will be conducted over 13 months.

The expected benefits can be major. The main benefit expected is the improvement of quality of life of the patients carrying the MEAVANTI breast prosthesis compared to those carrying the so-called standard prosthesis. A reduction in back and neck pain could also reduce the costs of patient management. In addition, this will demand referencing by the HAS of the custom-made prosthesis so that it is reimbursed in the same way as existing ones.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral mastectomy performed.
* Satisfactory healing
* Informed consent form signed.
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Elastomer type plastics or silicone allergy
* Contraindication to the use of the MEAVANTI or Standard external prosthesis: damaged or irritated skin in the area of application of the prosthesis
* Patient under the age of 18 years
* History of back problems (scoliosis)
* History of spine surgery
* Other cancer being treated,
* Dorsal hyperalgia
* Acute infectious episode (cellulitis, erysipelas, lymphangitis)
* Presence of subcutaneous osteosynthesis material with an external part at the level of the upper limb to be treated,
* Impossibility to comply with the constraints of the protocol,
* Pregnancy,
* Breast feeding
* Adult protected by law (tutelage, curators and safeguard of justice).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female with a breast cancer
Enrollment: 64 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Change in quality of life : emotional functioning | Change from baseline to 3 months
  Emotional dimension will be studied with items from 21 to 24 of EORTC Quality of Life Questionnaire QLQ-C30 (Generic Questionnaire) (Likert type with 4 choices from 1 = not at all to 4 = a lot)
Change in quality of life : social functioning | Change from baseline to 3 months
  Social dimension will be studied with items from 26 and 27 of EORTC Quality of Life Questionnaire QLQ-C30 (Generic Questionnaire) (Likert type with 4 choices from 1 = not at all to 4 = a lot)
Change in quality of life : body image | Change from baseline to 3 months
  Body image will be studied with items from 39 to 42 of EORTC Quality of Life Questionnaire BR23 Module (Breast Cancer Module) (Likert type with 4 choices from 1 = not at all to 4 = a lot)
Change in quality of life : sexual functioning | Change from baseline to 3 months
  Sexual functioning will be studied with items from 56 to 59 of EORTC Quality of Life Questionnaire BRECON 14 (Reconstruction module) (Likert type with 4 choices from 1 = not at all to 4 = a lot)
Change in quality of life : satisfaction breast cosmetic | Change from baseline to 3 months
  Satisfaction breast cosmetic will be studied with items from 60 to 65 of EORTC Quality of Life Questionnaire BRECON 14 (Reconstruction module) (Likert type with 4 choices from 1 = not at all to 4 = a lot)

SECONDARY OUTCOMES:
Visual satisfaction | 6 months
  Evaluation of the visual satisfaction associated with wearing of the external prosthesis by the self and the hetero-evaluation (from photos taken of the patient (face, profiles, ¾ with and without the prosthesis): carried out by a scale of judgment (Likert type with 5 choices from 1 = very satisfied to 5 = very unsatisfied) at 6 months.
Evaluation of pain | 3 months and 6 months
  Evaluation of pain by the analogical EVA scale 1 to 10, on the following 3 sites: back / shoulders / cervical at 3 monts and 6 months.
Comparative questionnaire | 6 months
  Comparative questionnaire "adhoc" between the 2 prostheses will be performed at 6 months (that is to say at the end of the study) targeting specific issues to the wearing of prostheses (previously used by the HAS for the referencing of silicone prostheses). This questionnaire consists of 14 questions, type Likert 5 points.
Collection of adverse events | 3 months and 6 months
  Adverse events will be recorded
Costs (consultations) | 1 month, 3 Months, 4 months and 6 months
  Costs for consultations will be raised
Costs (paramedical procedures) | 1 month, 3 Months, 4 months and 6 months
  Costs for paramedical procedures will be raised

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte VAYSSE, MCU-PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Rangueil, Toulouse, France, France

IPD SHARING:
Plan to Share IPD: No